CLINICAL TRIAL: NCT06296277
Title: Management of Mechanical Ventilation During Surgery: an International, Multicenter, and Observational Data Registry
Brief Title: Mechanical Ventilation in Surgical Patients
Acronym: MEET VENUS
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: University Of Perugia (Other); University of Chieti (Other); Medical University of Vienna (Other); The Netherlands Cancer Institute (Other); Monash University (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Prof Gianmaria Cammarota, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Other Study IDs: UPO#1!
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Surgery; Ventilator Lung; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intraoperative mechanical ventilation: Patients subjected to invasive mechanical ventilation (IMV) during general anesthesia for surgery
  Interventions: Other: Intraoperative mechanical ventilation for surgery

INTERVENTIONS:
Other: Intraoperative mechanical ventilation for surgery — Any IMV during general anesthesia for surgery

SUMMARY:
This is an investigator-initiated, international, multicenter, prospective, cross-sectional study that aims to 1) describe the incidence and types of postoperative pulmonary complications (PPCs), 2) describe patient demographics, baseline characteristics, and intraoperative ventilation management, 3) describe the occurrence of intraoperative adverse events (IAEs), and 4) their associations with PPCs, 5) assess the practice of intraoperative mechanical ventilation.

Patients will be eligible for participation if: 1) adult and 2) receiving intraoperative ventilation during general anesthesia for surgery. Patients receiving ventilation outside of an operating room as well as patients receiving intraoperative ventilation during extracorporeal life support will be excluded

DETAILED DESCRIPTION:
This is an investigator-initiated, international, multicenter, prospective, cross-sectional study The here proposed study aims to 1) describe the incidence and types of postoperative pulmonary complications (PPCs), 2) describe patient demographics, baseline characteristics, and intraoperative ventilation management, 3) describe the occurrence of intraoperative adverse events (IAEs), and 4) their associations with PPCs, 5) assess the practice of intraoperative mechanical ventilation.

Patients will be eligible for participation if: 1) adult and 2) receiving intraoperative ventilation during general anesthesia for surgery. Patients receiving ventilation outside of an operating room as well as patients receiving intraoperative ventilation during extracorporeal life support will be excluded.

The primary endpoint is to report the number of patients with PPCs occurring in the first 5 postoperative days. As secondary endpoint, the practice of mechanical ventilation in patients undergoing general anesthesia for surgery will be ascertained including key intraoperative ventilator characteristics and respiratory system mechanics. Other secondary endpoints will include: incidence and type of IAEs; postoperative complications other than PPCs in the first 5 postoperative days; intensive care unit (ICU) admission and length of stay, hospital length of stay, and hospital mortality on day 28.

Participating hospitals have the flexibility to choose a specific time period for data collection, but it is imperative that this process occurs within 8 weeks from receiving approval by the local Ethics Committee. Furthermore, each participating center will conduct data collection during a predetermined 7-day period. Local investigators will capture data in an electronic case recording form, including patient demographics and baseline characteristics, intraoperative ventilator settings and ventilation parameters, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults; and
* Receiving intraoperative IMV (via tracheal intubation, or supraglottic device ) during general anesthesia for surgery

Exclusion Criteria:

* Receiving intraoperative IMV outside of an operating room; and
* Receiving intraoperative IMV during extracorporeal life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to IMV during general anesthesia for surgery will be included in a consecutive manner
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications (PPCs) | within 5 days after surgery
  Incidence and type of PPCs

SECONDARY OUTCOMES:
Intraoperative adverse events (IAEs) | Intraoperatively
  Incidence and type of IAEs
Intraoperative mechanical ventilation practice | Intraoperatively
  Mechanical ventilation settings in patients undergoing general anesthesia for surgery
Postoperative clinical outcome | Postoperatively, on day 28 following surgery
  Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Gianmaria Cammarota, Prof, Principal Investigator — Università degli Studi del Piemonte Orientale; Rachele Simonte, MD, Study Director — University Of Perugia; Edoardo M De Robertis, Prof, Study Director — University Of Perugia; Sabrine N.T. Hemmes, MD, Study Director — Department of Anesthesiology The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, The Netherlands; Marcus J Schultz, Prof, Study Director — Department of Anaesthesia, General Intensive Care & Pain Management, Medical University of Vienna; Salvatore M Maggiore, Prof, Study Chair — Department of Anesthesiology and Intensive Care, Ospedale SS Annunziata & Department of Innovative Technologies in Medicine and Odonto-stomatology, Università Gabriele D'Annunzio di Chieti-Pescara, Chieti, Italy; Ary Serpa Neto, Prof, Study Director — Australian and New Zealand Intensive Care Research Centre (ANZIC-RC), School of Public Health and Preventive Medicine, Monash University, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Undecided